CLINICAL TRIAL: NCT03421457
Title: A Multicenter, Randomized, Prospective, Controlled Study Comparing Uterine Preserving Laparoscopic Lateral Suspension With Mesh Versus Laparoscopic Sacrocervicopexy in the Treatment of Uterine Prolapse: A Randomized Controlled Trial
Brief Title: Laparoscopic Lateral Suspension With Mesh & Sacrocervicopexy for the Treatment of Uterine Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, MURAT YASSA, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCTPOPS
Record Dates: First submitted 2018-01-21; First posted 2018-02-05 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse; Pelvic Floor Prolapse
Keywords: Pelvic Organ Prolapse; Translabial ultrasound; Transperineal ultrasound; Lateral Mesh Suspension; Descensus uteri; Laparoscopic pelvic organ prolapse repair; Uterus preserving; hysteropexy; uterine-preserving; fertility-sparing; sacropexy; cervicopexy; sacrocervicopexy; sacrohysteropexy; mesh prolapse surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider will be blind to the operation type. Outcomes will be assessed by a gynecologist who will be blind to the operation type, indications and complications. Assessor has wide experience in urogynecological sonography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral suspension (Experimental): "Uterus-preserving Laparoscopic lateral suspension with mesh" technique will be performed in this arm.
  Interventions: Procedure: Uterus-preserving laparoscopic lateral suspension with mesh
- Sacrocervicopexy (Experimental): "Uterus-preserving Laparoscopic sacrocervicopexy with mesh" technique will be performed in this arm.
  Interventions: Procedure: Uterus-preserving laparoscopic sacrocervicopexy with mesh

INTERVENTIONS:
Procedure: Uterus-preserving laparoscopic lateral suspension with mesh — V-shaped 2cm wide and 25cm length mesh strip is prepared from a 30x30cm Prolene mesh (Ethicon J&J).Deep dissection of the uterovesical space is performed.Cutaneous incisions are bilaterally made 3-4 cm superoposterior to the anterosuperior iliac spine.A grasper is introduced retroperitoneally through the sub-peritoneum holding the beginning part of mesh until reaching the vesicovaginal space in an oblique route rather than transverse.Round ligament is lifted upward and tunnel is practiced horizontally.Assistant grasper catches the distal mesh and pulls out through the opposite subperitoneal tunnel.Corner of mesh is fixed to the pubocervical fascia,uterine cervix and isthmus with Absorba-Tack™(Covidien, Mansfield,USA).Tension-free lateral mesh suspension is achieved at the desired level.
  Arms: Lateral suspension
Procedure: Uterus-preserving laparoscopic sacrocervicopexy with mesh — The peritoneum over the sacral promontory is incised until the anterior longitudinal ligament is reached and ureters are identified. Peritoneal relaxing incision is made medial to the right ureter, down into the pelvis, posterior to the cervix and rectovaginal fascia, laterally to the rectum. The arm of the mesh is sutured to the posterior cervix by 2.0 prolene and fixated to the sacral promontory by either Tacker (Covidien) and/or 2.0 prolene as tension-free. Complete peritonisation of the mesh is performed.
  Arms: Sacrocervicopexy

SUMMARY:
This study is aimed to compare the efficiency of two uterus-preserving laparoscopic methods to treat uterine prolapse in a randomized controlled trial. Laparoscopic lateral suspension with mesh (LLSM) will be compared with laparoscopic sacrohysteropexy (LS). Both procedures are known as sufficient uterus preserving methods. LLSM was introduced to be an alternative to others with avoiding dissection of promontory and therefore being safer, faster and feasible technique.

DETAILED DESCRIPTION:
Patient with uterine prolapse can participate in this study. A total of 44 women will be included. At random 22 patients undergo laparoscopic lateral suspension with mesh operation and 22 patients undergo laparoscopic sacrohysteropexy operation. Evaluation will take place during the surgery, at the postoperative visit after 4 weeks, 6th months and 12th months. Quality of life, degree of vaginal prolapse, safety, operation time and complications will be evaluated.

Subjective assessments will include Female Sexual Function Index (FSFI), Michigan Incontinence Severity Index (M-ISI), Prolapse Quality of Life questionnaire (PQoL), Pelvic Organ Prolapse Symptom Score (POP-SS) and Visual Analog Score (VAS).

Objective assessments will include routine gynecologic sonography, Pelvic Organ Prolapse Quantification System (POP-Q) and pelvic floor biometry measured by transperineal sonography.

Transperineal sonography will include those measurements:

Urethral rotation, Pelvic organ descent, Hiatal Diameter and the Anatomical localization of apex.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* > Symptomatic prolapse of central compartment with a Pelvic Organ Prolapse Quantitative (POP-Q) stage 2 associated or not with anterior or posterior compartment prolapse.
* Patients who are not comfortable with using or refusing pessary
* Wish to preserve the uterus

Exclusion Criteria:

* Any cue for gynecologic oncological condition
* Patients who approves Le Fort colpocleisis among who does not have any sexual intercourse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline POP-Q measurements (mm) at 12th month. | 12 months for each participant
  Prolapse degree; Point Ba/C/Bp

SECONDARY OUTCOMES:
Subjective Success - Change from baseline Female Sexual Function Index (FSFI) to measure sexual dysfunction at 12th month. | 12 months for each participant
  Validated into Turkish language form will be used to compare preoperative and postoperative period. The FSFI is a multiple-trait scoring, self-report document used to assess female sexual function. It consists of 19 items that encompass six separate domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The maximum score is 36 points and the minimum score is 2 points. After completion of the questionnaire, the total SF score was calculated as follows: no sexual dysfunction (SD) (≥ 30 points) , mild SD (between <29 and > 23 points), and severe SD (≤ 22 points).
Subjective Success - Change from baseline Michigan Incontinence Severity Index (M-ISI) to measure urinary incontinence at 12th month. | 12 months for each participant
  Validated into Turkish language form will be used to compare preoperative and postoperative period. It has ten items, consisting of a total M-ISI domain (the sum of items 1-8) and a distinct Bother domain (the sum of items 9 and 10). The total M-ISI score consists of three subdomains (items 1-3 for stress urinary incontinence [SUI], items 4-6 for UUI, and items 7 and 8 for PU). The responses for each item range from 0 to 4 on a Likert-type scale, with higher values representing greater symptoms and greater bother. The total M-ISI domain ranges from 0 to 32, the Bother domain ranges from 0 to 8, the SUI and UUI subdomains range from 0 to 12, and the PU subdomain ranges from 0 to 8. Total domain and subdomain scores are obtained by simply adding the respective answers. The minimally important difference has been determined for the following domains/subdomains: total M-ISI (4 points), SUI (2 points), UUI (2 points), and PU (1 point).
Subjective Success - Change from baseline Prolapse Quality of Life questionnaire (PQoL) to measure quality of life according to pelvic organ prolapse at 12th month. | 12 months for each participant
  Validated into Turkish language form will be used to compare preoperative and postoperative period. he questionnaire included 20 questions grouped in sections (domains) related to a particular aspect of quality of life. A total of nine domains covering general health, prolapse impact, role limitations, physical and social limitations, personal relationships, emotional problems, sleep/energy disturbance as well as severity symptoms measurements were defined. Questions regarding bladder, bowel and sexual function were also separately included and validated for reproducibility and internal consistency. Responses ranged from 'none/not at all', through 'slightly/a little' and 'moderately' to 'a lot' to produce a four-point scoring system for each item. Scores in each domain ranged between 0 and 100 with a high total score indicating a greater impairment of quality of life.
Subjective Success - Change from baseline Pelvic Organ Prolapse Symptom Score (POP-SS) to measure quality of life according to pelvic organ prolapse at 12th month. | 12 months for each participant
  Validated into Turkish language form will be used to compare preoperative and postoperative period. Total range scores: 28 (min:0, max:28). Higher values represent a worse outcome.
Subjective Success - Change from baseline Visual Analog Score (VAS) for pain at 12th month. | 12 months for each participant
  Participant describes the pain related to the mesh. The respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain with a format of a horizontal bar.
Change from baseline Pelvic Hiatus measurements (mm) at 12th month. | 12 months for each participant
  Anteroposterior hiatal length (mm)
Change from baseline Pelvic biometry measurements at 12th month. | 12 months for each participant
  Prolapse degree over symphysis pubis (mm) Anterior compartment over 10mm, Posterior compartment over 15 mm are clinically relevant
Change from baseline bladder neck mobility measurements at 12th month. | 12 months for each participant
  Urethral rotation (degree) between rest and valsalva maneuver states
Failure (%) | 12 months for each participant
  Failure is defined by any recurrence of prolapse, mesh erosion and need for additional surgery
Complications | 12 months for each participant
  Perioperative and postoperative complications including Severe bleeding, hematoma, bladder injury, bowel injury, ureter injury, vascular injury, nerve injury, abscess, lower urinary tract infections, mesh extrusion, mesh exposure, prolapse recurrence, De novo SUI/OAB, dyspareunia, pelvic pain
Operation time | Operation time will noted for each participant at the same day of the operation. Operation time will be determined with using a chronometer,from the time of first skin incision until the suturing the skin of the trocar entry, assessed up to 52 weeks.
  Duration of the operation between the first skin incision and suturing the skin of the trocar entries

CONTACTS AND LOCATIONS:
Overall Officials: Niyazi Tug, As.Prof., Study Director — Chief of the Department
Locations (2):
- Turkey (Türkiye) (2):
  - Fatih Sultan Mehmet Training and Research Hospital, Sancaktepe Campus, Istanbul, Sancaktepe
  - Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Sisli

IPD SHARING:
Plan to Share IPD: No
Study Protocol

REFERENCES:
- [Background] Veit-Rubin N, Dubuisson JB, Gayet-Ageron A, Lange S, Eperon I, Dubuisson J. Patient satisfaction after laparoscopic lateral suspension with mesh for pelvic organ prolapse: outcome report of a continuous series of 417 patients. Int Urogynecol J. 2017 Nov;28(11):1685-1693. doi: 10.1007/s00192-017-3327-2. Epub 2017 Apr 17. PMID 28417156